CLINICAL TRIAL: NCT06767306
Title: A Phase II, Multicentre, Non-Comparative, Randomised Controlled Trial of Stereotactic Ablative Body Radiotherapy and Immunotherapy Versus Immunotherapy Alone in Patients With Treatment Naïve Oligometastatic Extracranial Melanoma
Brief Title: Stereotactic Ablative Radiotherapy (XRT) and Immunotherapy for Oligometastatic Extracranial Melanoma
Acronym: AXIOM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIA2024/508
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Melanoma Metastatic
Keywords: SABR; stereotactic body radiotherapy; Stereotactic Ablative Body Radiotherapy; SABRT; Immunotherapy; Immune Checkpoint Inhibitors; Oligometastases; Extracranial; Quality of life; Biomarkers
MeSH Terms: interventions — Radiosurgery; Immunotherapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Open label, 2-arm parallel group, non-comparative, randomised (2:1 ratio) controlled, trial with stratification by:
  * Liver metastasis vs no liver metastasis
  * Baseline LDH: normal vs elevated
  * Immunotherapy agents: anti-PD-1 alone vs anti-PD-1 combination with anti-CTLA-4 or anti-LAG-3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Concurrent stereotactic body radiotherapy + Immune checkpoint inhibitor(s) (Experimental): Concurrent stereotactic body radiotherapy (SBRT) with standard of care immune checkpoint inhibitor(s) (ICI).
  Patients will receive a minimum SBRT biologically effective dose (BED) of 48Gy10 to all sites of metastatic disease between cycle 1 and cycle 3 of immunotherapy. The interval between cycles 1 and 3 will depend on the prescribed immunotherapy regimen that is standard of care at each participating site.
  Standard of care 1st line immunotherapy, as decided by the treating clinician and in accordance with the current listing on the Australian Register of Therapeutic Goods (ARTG) or applicable international regulatory agency will be administered concurrently
- Arm B: Immune checkpoint inhibitor(s) (Active Comparator): Immunotherapy alone
  Standard of care 1st line immunotherapy, as decided by the treating clinician and in accordance with the current listing on the Australian Register of Therapeutic Goods (ARTG) or applicable international regulatory agency will be administered alone.
  Interventions: Drug: Immunotherapy alone

INTERVENTIONS:
Other: Stereotactic Body Radiotherapy (extracranial) concurrent with Immunotherapy — Radiotherapy A minimum SBRT biologically effective dose (BED) of 48Gy10 to all sites of extracranial metastatic disease should be administered between cycle 1 and cycle 3 of standard of care immunotherapy.
  Immunotherapy All patients will receive standard of care 1st line immunotherapy as decided by the treating clinician and in accordance with the current listing on the Australian Register of Therapeutic Goods (ARTG) or applicable international regulatory agency.
  Other Names:
  Immune checkpoint inhibitor Standard of care immunotherapy First line treatment
Drug: Immunotherapy alone — All patients will receive standard of care 1st line immunotherapy as decided by the treating clinician and in accordance with the current listing on the Australian Register of Therapeutic Goods (ARTG) or applicable international regulatory agency.
  Other Names: Immune checkpoint inhibitor; Standard of care immunotherapy; First line treatment
  Arms: Arm B: Immune checkpoint inhibitor(s)

SUMMARY:
The purpose of this research is to evaluate the addition of radiotherapy to the standard immunotherapy drugs that are given to patients with advanced or metastatic melanoma that has spread to other parts of the body. Radiotherapy uses x-rays to target and kill melanoma cells and immunotherapy works by activating the body's own immune system to seek out and ﬁght melanoma cells. Both of these treatments are commonly given to patients with advanced melanoma and other cancers. Both treatments are usually given separately but can also be given together. The aim of this research is to find out if giving radiotherapy and immunotherapy together is better than giving immunotherapy alone.

The type of radiotherapy to be used in this project is known as 'stereotactic' body radiotherapy or SBRT (also known as stereotactic body ablative radiotherapy, SABR). SBRT targets the radiation very precisely at the metastatic deposits in the body. This method protects the healthy areas near the melanoma. SBRT works by delivering a high dose of radiation precisely to the areas of melanoma which causes the melanoma cells to break apart and eventually die. SBRT is given in 'fractions' which means the high dose is given in small measures over several days, depending on the number and size of metastases.

DETAILED DESCRIPTION:
One of the promising treatment combinations for metastatic melanoma is the use of radiotherapy with immune checkpoint inhibitors. There have been multiple reports of the synergy between radiation and immunotherapy in preclinical studies and early phase clinical trials. This combination improves response rates compared to immunotherapy alone and without worsening the toxicity associated with each agent alone. Radiation has the potential to convert tumours considered immunologically "cold" into "warm" through the combination of three processes: 1) Changes in the balance of cytokines by increasing the production of immunostimulatory cytokines which overcome the immunosuppressive tumour microenvironment, 2) Recruitment, of antigen-presenting cells and immune effector cells in the tumour microenvironment, 3) Positive regulation of antigen expression, antigen processing, histocompatibility molecules, and costimulatory signals, thereby increasing tumour immunogenicity.

There is a significant body of data to suggest a reproducible clinical benefit can be achieved when stereotactic body radiotherapy (SBRT) is used with immunotherapy in a tightly sequenced treatment combination, in contrast to independently timed use of either treatment alone, for the management of a variety of malignancies. In metastatic non-small cell lung cancer, a pooled analysis of two randomised trials showed that the addition of radiotherapy improved the out-of-field response rate, progression-free survival, and the overall survival. In the Stereotactic Ablative Radiotherapy for Comprehensive Treatment of Oligometastatic Tumors trial (SABR-COMET - NCT01446744) of 1-5 oligo metastases in all tumour histologies, the 8-year overall survival was 27.2% in the experimental SBRT arm versus 13.6% in the palliative radiotherapy control arm (with the goal of alleviating symptoms) (hazard ratio, 0.50; 95% confidence interval, 0.30-0.84; P = 0.008). The eight-year progression free survival estimates were 21.3% versus 0.0%, respectively (hazard ratio, 0.45; 95% confidence interval, 0.28-0.72; P <0.001) (Harrow, Palma et al. 2022). There are two ongoing phase 3 randomised trials of SABR with standard of care (palliative radiotherapy with or without systemic anti-cancer therapy) vs standard of care alone for patients with 1-3 solid cancer metastases (SABR-COMET 3) and 4-10 metastases (SABR- COMET 10).

At present, patients with metastatic melanoma receive various treatment modalities in different combinations and sequencing, including a drug alone approach, palliative radiotherapy for symptom control, SBRT to persistent disease as salvage therapy if all or some metastases do not respond to initial drug therapy, and surgery. There is an ongoing randomised trial examining the role of upfront stereotactic radiosurgery to asymptomatic melanoma brain metastases in patients receiving concurrent combination of ipilimumab and nivolumab (Clinical Trials.gov Identifier: NCT03340129). However, there is no prospective randomised trial on the role of SBRT with immunotherapy in patients with extracranial melanoma oligometastases.

The AXIOM trial seeks to determine the role of upfront SBRT in patients with 1-5 extracranial melanoma oligometastases treated with concurrent immunotherapy. The efficacy of immunotherapy in this patient population is well established and therefore this randomised controlled study design is non-comparable with the control group. The randomisation ratio of 2:1 will provide more information on the response and safety of SBRT and immunotherapy, whilst limiting the number of patients randomised to the 'control' group, in order to provide minimum but contemporary immunotherapy efficacy and safety data.

The hypothesis is that for patients with extracranial melanoma oligometastases, concurrent stereotactic body radiotherapy with immunotherapy is safe and prolongs survival through enhanced anti-tumour immunity due to the potential synergy of the combination therapies, than immunotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients, age 18 or older
* Willing to provide signed informed consent
* Life expectancy > 6 months
* First presentation of AJCC Stage IV (any N, M1a, M1b, M1c), histologically confirmed cutaneous, acral or unknown primary melanoma with one to five extracranial metastases detected on CT and whole body PET-CT, and considered unresectable
* A primary lesion and / or up to 4 in-transit metastases(is) (ITM) in addition to distant metastases(is) are permitted and will be counted in the maximum number of permitted baseline lesions
* Prior surgery for symptomatic disease (e.g. small bowel obstruction) for this first presentation of Stage IV melanoma is permitted, provided the total number of remaining extracranial metastases is ≤ 5 (NOT including the resected lesion). No more than one excised metastatic lesion is permitted
* At least one metastasis should be measurable as a target lesion per RECIST version 1.1
* No evidence of cerebral metastases on MRI brain (CT brain is acceptable if there is contraindication to MRI)
* All lesions can be treated with a minimum SBRT biologically effective dose (BED) of 48Gy
* Able to tolerate treatment with immunotherapy as determined by the medical oncologist
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of randomisation

Exclusion Criteria:

* Ocular or mucosal melanoma
* Serious or unstable medical co-morbidities or other conditions that could interfere with the patient's safety, consent, or compliance
* Patients for whom there is a definite and immediate indication for radiotherapy (e.g., spinal cord compression, rapidly progressing disease associated with clinical signs and symptoms)
* Prior radiotherapy for Stage IV disease (prior adjuvant radiotherapy to primary site or nodal field (Stage I-III disease) is permitted, however adjuvant-treated sites must not be included in the baseline lesions
* Inability to treat all disease sites with SBRT as determined by radiation oncologist
* Prior systemic drug therapy for melanoma, unless given in the neoadjuvant or adjuvant setting for Stage I-III disease
* Any contraindication to the planned standard of care immunotherapy regimen per regulatory approved product information
* For patients with liver metastases - moderate/severe liver dysfunction
* A known history of another malignancy or concurrent malignancy unless the patient is disease-free for a minimum of 1 year, is completely treated and is at low risk of recurrence
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2033-04-01 (Estimated); Study Completion 2033-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Proportion of patients alive at 6 months 1, 2, 3 and 5 years from the time of randomization

SECONDARY OUTCOMES:
Overall progression-free survival | 5 years
  Proportion of patients alive and with no evidence of disease progression or new melanoma lesions as assessed by RECIST 1.1 criteria
Progression-free survival related to new lesions only | 5 years
  Proportion of patients alive and with no evidence of new melanoma lesions as assessed by RECIST 1.1 criteria
Overall response rate | 5 years
  Overall response rate from the time of randomization to the best response as assessed by RECIST 1.1
Local control of the initial oligometastases | 5 years
  The proportion of patients with local control of all baseline metastases: complete response, partial response or stable disease) as assessed per RECIST 1.1 criteria
Safety and tolerability of each treatment arm and study procedures | 5 years
  Proportion of patients with adverse events related to SBRT alone, combined SBRT and immunotherapy, immunotherapy-related Suspected Unexpected Serious Adverse Reaction (SUSAR), or related to study specific procedures with causality determined by the investigator and described per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Only AEs greater than CTCAE grade 1 will be recorded.
The requirement for immunosuppressive agents to treat adverse events | 5 years
  Proportion of patients receiving corticosteroids or other immunosuppressive agents to treat each adverse event including duration and maximum dose.
Patient reported quality of life | 5 years
  The mean change from baseline quality of life scores [EuroQol Group Association ED-5Q-5L and European Organisation for Research and Treatment of Cancer QLQ-C30] from randomization to best and lowest scores for each instrument.
Salvage radiotherapy in the immunotherapy alone arm | 5 years
  The incidence of salvage radiotherapy for symptomatic control or progressing baseline lesions or new metastasis(es) in the immunotherapy arm.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hong, Study Chair — Melanoma Institute Australia
Locations (4):
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hong AM, Wang T, Carlino MS, Lo SN, Menzies AM, da Silva IP, Long GV. Study protocol of a randomised phase II trial of concurrent stereotactic body radiotherapy with immunotherapy versus immunotherapy alone in patients with 1-5 extracranial melanoma oligometastases (AXIOM). BMC Cancer. 2025 Oct 21;25(1):1615. doi: 10.1186/s12885-025-15066-z. PMID 41120904